CLINICAL TRIAL: NCT03840824
Title: Blood Spot Self-administered Test and Assay
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 812735
Record Dates: First submitted 2015-03-17; First posted 2019-02-15 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Dysfunction; Endocrine; Effects of Chemotherapy; Premature Ovarian Failure
Keywords: healthy; premenopausal; postmenarchal; chemotherapy; alkylating agent; alkylator; high dose cancer therapy; low dose cancer therapy
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Cancer Survivor: Pre-menopausal women who are cancer survivors ages 18-45 years with normal menstrual cycles.
- Similar aged healthy controls: Pre-menopausal, healthy women ages 18-45 years with normal menstrual cycles
- Late Reproductive Age: Pre-menopausal, healthy women of late reproductive age

SUMMARY:
The current study will compare hormone levels of AMH, FSH and inhibin B in blood specimens collected by venipuncture and fingerstick in a sample of pre-menopausal women ages 18-45 years with normal menstrual cycles.

DETAILED DESCRIPTION:
Recent advances in cancer diagnosis and treatment have led to greater survival rates in patients with malignancies. However, these life-saving treatments, especially alkylating agents, often lead to premature ovarian failure, infertility and related long-term health problems. It is difficult to predict whether, and the extent to which, patients will experience these problems. There are no early clinical signs of decreased fertility potential; even young women who maintain cyclic menses after therapy are at high risk of infertility, early menopause and related health problems. Preliminary studies suggest that several surrogate measures of fertility potential are different in cancer survivors compared with controls. These include follicle stimulating hormone (FSH), estradiol, anti-mullerian hormone (AMH) and inhibin B. Large longitudinal studies are needed to validate these measures with gold standard outcomes such as pregnancy rates, pregnancy outcomes and time to menopause. The main impediment to assessing the value of these markers and generating data that is useful to cancer survivors is the need for frequent and timed blood samples.

Daily or frequent trips to the clinical center are not practical and reduce the compliance of even the most motivated patients. The hypothesis that will be tested by this study is that blood spot assays can be developed that provide robust, personalized data for surrogate markers of reproductive function which can be used to assess reproductive potential in women; furthermore, bloodspots collected at home are an acceptable method for reproductive hormone measurement in women with and without a history of cancer. The current study will compare hormone levels of AMH, FSH and inhibin B in blood specimens collected by venipuncture and fingerstick in a sample of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Adult females
* Age between 18-45 years
* Premenopausal (defined as menses in the past 12 months)
* Postmenarchal
* Presence of an intact uterus and two ovaries
* Ability and willingness to comply with study protocol

Exclusion Criteria:

* Pregnancy within the previous 3 months
* Lactation within the previous 3 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target population is 80 pre-menopausal women ages 18-45 years with normal menstrual cycles:
  Aim 1: Total 80 subjects:
  * 30 cancer survivors
  * 30 similar aged healthy controls
  * 20 late reproductive aged women
  Aim 2: Subset of 60 subjects:
  * 30 cancer survivors
  * 30 similar aged healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2016-06 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
AMH pg/mL in dried bloodspot vs serum samples | Day 1
  Serum AMH ELISA assay results will be compared to capillary blood sample AMH collected on filter paper and dried. Recovery of spiked ligands, sensitivity and specificity of the assays will be also assessed.

SECONDARY OUTCOMES:
Adequacy of subject's self-collected bloodspot sample vs. sample collected in clinic | Day 1
  A capillary blood sample from a finger-prick is applied to Whatman #903 filter paper, allowed to dry at room temperature for at least 4 hours, and then stored until analysis in the laboratory. Subjects willing to conduct a finger stick at home will collect an additional dried blood spot sample for secondary outcome measures. At home blood spot cards will be compared to those obtained in the office to determine adequacy of collection.
Measures of user acceptability through subject report/feedback | Day 1
  Ease of use data reported by subject survey will be summarized to determine the overall acceptability of bloodspot collection and the potential for at- home use
AMH pg/mL in cancer survivors vs. healthy control cohorts | Day 1
  AMH in dried blood spots vs. serum collected during the early follicular phase in 30 cancer survivors (15 exposed to low dose cancer therapy, 15 exposed to high dose cancer therapy) and 30 healthy similar aged controls will be compared using tests and multivariable linear regression
FSH (mIU/mL) in dried bloodspot vs serum samples | Day 1
  Serum FSH ELISA assay results will be compared to FSH in a dried capillary blood sample applied to filter paper. Recovery of spiked ligands and sensitivity and specificity of the assays will be assessed.
Inhibin B (pg/ml) in dried bloodspot vs serum samples | Day 1
  Serum Inhibin B ELISA assay results will be compared to capillary blood sample Inhibin B collected on filter paper and dried. Recovery of spiked ligands and sensitivity and specificity of the assays will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Clarisa Gracia, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Reproductive Research Unit, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] McDade TW, Woodruff TK, Huang YY, Funk WE, Prewitt M, Kondapalli L, Gracia CR. Quantification of anti-Mullerian hormone (AMH) in dried blood spots: validation of a minimally invasive method for assessing ovarian reserve. Hum Reprod. 2012 Aug;27(8):2503-8. doi: 10.1093/humrep/des194. Epub 2012 Jun 6. PMID 22674205